CLINICAL TRIAL: NCT01402921
Title: Efficacy on Volume Reduction and Tolerance of Progressiv' Medical Compressive Therapy (MCT) V0322 BC in Patients With Chronic Venous Oedema. International, Multicentric, Randomised, Controlled, Double Blind Study, in Two Parallel Groups v0322 bc Versus Placebo
Brief Title: Efficacy on Volume Reduction and Tolerance of Progressiv' Medical Compressive Therapy (MCT) V0322 BC in Patients With Chronic Venous Oedema
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: V00322 BC 402
Record Dates: First submitted 2011-07-13; First posted 2011-07-26 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Venous Insufficiency (CVI)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elastic Medical Compressive Therapy (Experimental): V0322BC verum medical compressive therapy is a progressive compressive sock with:
  * ankle pressure: 10 mmHg
  * calf pressure : 23 mmHg
  Interventions: Device: V0322 BC
- Placebo (Placebo Comparator): V0322BC placebo medical compressive therapy is a progressive compressive sock with:
  * ankle pressure: <5 mmHg
  * calf pressure : <7 mmHg
  Interventions: Device: V0322 BC

INTERVENTIONS:
Device: V0322 BC — * Stocking Elastic MCT is a widely recognized and the consensus-approved treatment for chronic venous insufficiency (CVI).Efficacy evidence level is often insufficient (grade B or C), or based on studies carried prior to CEAP classification (2004).
  * The medical device is defined by the following parameters: ankle pressure(10 mmHg)and calf pressure (23 mmHg)
  * 3 months duration daily treatment

SUMMARY:
Elastic MCT is a widely recognized and the consensus-approved treatment for chronic venous insufficiency (CVI).Efficacy evidence level is often insufficient (grade B or C), or based on studies carried prior to CEAP classification (2004). Item C3 of this classification relates to patients suffering from chronic venous disease and permanent oedema. Literature mentions only one study in which volume reduction in venous-induced oedema was primary endpoint. Indeed, 240 patients showed a 46.7 ± 8.2 ml reduction (SEM) after 12 weeks with a Class 2 compression sock (15-20 mm Hg at ankle). Volume is an accurate and reproducible quantitative measure considered nowadays as being gold standard when objectifying oedema variation. It is therefore particularly relevant in a C3-patient trial (CEAP classification).

The main objective of the current study is to evaluate the clinical effect of Progressiv' MCT on volume reduction in permanent CVI-oedema after 3 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Permanent chronic oedema of venous origin (C3 based on CEAP classification) confirmed by Doppler or Duplex ultrasound examination with reflux and/or obstruction on superficial, deep or perforator veins
* Pitting oedema
* Have given and signed written informed consent
* Registered with or benefiting from health insurance (Mandatory for France)

Exclusion Criteria:

* Use of compression therapy in the last 5 days before inclusion
* Common contraindications for MCT (arteriopathy, decompensated heart failure, infectious dermatitis
* Isolated lipoedema
* Isolated lymphoedema (Kaposi- Stemmer sign
* Severe systemic disease (heart failure, renal failure, hepatic failure, thyroid dysfunction untreated, malnutrition with hypo-proteinemia …)
* Known hypersensitivity to any component of MCT
* Important limitation of ankle movement requiring a specific therapy
* Following treatment initiated or dose-modified 1 month prior to inclusion: NSAID, corticosteroids, calcium blockers, ACE inhibitors, Angiotensin II inhibitors, vasoconstrictors or vasodilators
* Hormonal treatment initiated or dose-modified 1 month prior to inclusion
* Diuretic and/or phlebotonic treatment initiated or dose-modified 1 month prior to inclusion
* Pregnancy, breast feeding, planning to become pregnant, or not using any form of contraception
* Patient linguistically or psychologically unable to understand the information given or who refuses to give his/her consent in writing
* Participation in another clinical trial
* Deprived of liberty for administrative, medical and legal reasons
* May not be compliant with the constraints imposed by the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Volume reduction of the target leg presenting the most important initial volume (by Volumetry using water displacement) | Day 90
  The main criterion is defined as the target leg volume reduction of chronic venous oedema measured by volumetry method with water displacement at 3 months

SECONDARY OUTCOMES:
Functional symptoms by VAS (pain, heaviness) at each visit by the patient. | 0-Day 7-Day 30 and Day 90
Quality of life. SQOR-V and ABC-V (FARDEAU) score | 0-Day 7-Day 30 and Day 90
Body weight variation | 0-Day 7-Day 30 and Day 90
Suprafacial Thickness Measured Duplex measurement | 0-Day 7-Day 30 and Day 90
Assessment of local tolerance (examination of the skin) and safety (general clinical examination and reported adverse events) | Day 7-Day 30 and Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalo-Universitaire Grenoble, Grenoble, Isère, France